CLINICAL TRIAL: NCT06731335
Title: Psilocybin for Enhanced Analgesia in Chronic nEuropathic PAIN
Acronym: PEACE-PAIN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P-005
Record Dates: First submitted 2024-11-28; First posted 2024-12-12 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Chronic Neuropathic Pain; Pain Management
Keywords: chronic pain; neuropathic pain; psychodelics; psilocybin; chronic neuropathic pain
MeSH Terms: conditions — Agnosia; Chronic Pain; Neuralgia | interventions — Psilocybin; Psychotherapy

STUDY DESIGN:
Intervention Model Description: Feasibility trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm with Psilocybin (Experimental): Intervention Arm with Psilocybin 25 mg single dose PO + psychological support
  Interventions: Drug: Psilocybin
- Placebo (Placebo Comparator): Placebo (Active) Dextromethorphan 400 mg single dose PO + psychological support
  Interventions: Drug: Active Placebo

INTERVENTIONS:
Drug: Psilocybin — PSILOCYBIN (PEX010) 25 mg PO single dose
  Other Names: Psychotherapy
  Arms: Intervention Arm with Psilocybin
Drug: Active Placebo — Dextromethorphan 400 mg PO single dose
  Other Names: Psychotherapy
  Arms: Placebo

SUMMARY:
This is a feasibility study to examine the use of use of Psilocybin (magic mushrooms) to alleviate pain in chronic neuropathic pain.

While theoretical mechanisms demonstrate promise, there is no clinical evidence. This vacuum of clinical evidence has been occupied by a "psychedelic hype bubble" with media communications touting psychedelics as a 'miracle cures'. The mismatch between evidence and perception creates an urgent need for RCT to fill this significant gap. This trial aims to address this gap by conducting a pilot trial assessing the feasibility, tolerability, and preliminary efficacy of psilocybin for chronic neuropathic pain to inform a future larger, multi-centre study.

The purpose is to conduct a randomized control double-blinded trial of psilocybin and active placebo (dextromethorphan).

At this time, the aim of the trial is to recruit 30 participants from St. Michael's Hospital, to learn whether it will be feasible to plan a larger study in the future.

DETAILED DESCRIPTION:
Brief title PEACE-PAIN Trial Indication Adult patients suffering from chronic neuropathic pain Condition(s) of focus of study Moderate-to-severe chronic neuropathic pain Number of participants 30 Primary outcome Feasibility (recruitment success, consent rate, adherence, patient withdrawal, missing data, adverse outcomes) Secondary outcome Change in pain intensity and pain interference Study design Study type: An intervention trial Allocation: Randomized Intervention model: 2-Arm Parallel Group Primary purpose: Feasibility Phase: Phase II Masking Participants, all study team including outcome assessors

Test Products, Dose, and Mode of Administration Treatment arm: Psilocybin 25mg + placebo PO single dose plus psychological support Placebo arm: Dextromethorphan 400mg PO single dose plus psychological support

Follow-Up Days: 1, 7, 14, 30, and 90

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Diagnosis of chronic neuropathic pain as determined by a pain specialist
* Moderate-to-severe neuropathic pain determined by Patient Reported Outcomes Measurement Information System (PROMIS)
* Previous trials of at least two medications recommended in the Canadian consensus guidelines on the management of neuropathic pain with no self-reported meaningful improvement in symptoms
* Sufficient command of English to participate in psychotherapy
* For participants of childbearing potential, use of a highly effective or double-barrier methods of contraception.

Exclusion Criteria:

* History of Dextromethorphan addiction or abuse.
* Enzyme CYP2D6 deficient as shown on the pharmacogenetic test.
* Underlying psychiatric conditions: lifetime or family history of a primary psychotic disorder, bipolar disorder, borderline personality disorder, paranoid personality disorder, current suicidal ideation, and substance use disorder within the past 12 months as assessed by history and confirmed by the Mini International Neuropsychiatric Interview (MINI)
* Medications that interact with study drugs
* Medical condition that is unstable or inadequately controlled, including cardiovascular disease, liver disease, or end-stage renal disease
* Previous lifetime use of a serotonergic psychedelic drug
* Nursing or pregnant women.
* Any other clinically significant medical illness that, in the opinion of the investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if they take part in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility to recruit 30 participants into a trial of psilocybin and active placebo to prepare for a larger multicentre trial | 18 months
  Recruitment rate and withdrawal rate (Acceptability and feasibility study)

SECONDARY OUTCOMES:
Change in pain intensity from baseline to one month after interventions | one month
  Patient-Reported Outcomes Measurement Information System Pain Interference, PROMIS Pain Intensity, Pain intensity scale- 0 to 10 (The higher the number the higher the pain intensity)
Change in pain interference from baseline to one month after interventions | one month
  Patient-Reported Outcomes Measurement Information System Pain Interference, PROMIS 6 a. Pain Interference, Pain interference scale- 6 items, 5 Likert scale (the higher the score the higher the interference from pain)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital. Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No individual participant data has been planned to be shared with other researchers at this point, since this is a feasibility study with only 30 participants

REFERENCES:
- [Background] Griffiths RR, Johnson MW, Richards WA, Richards BD, McCann U, Jesse R. Psilocybin occasioned mystical-type experiences: immediate and persisting dose-related effects. Psychopharmacology (Berl). 2011 Dec;218(4):649-65. doi: 10.1007/s00213-011-2358-5. Epub 2011 Jun 15. PMID 21674151
- [Background] Carbonaro TM, Bradstreet MP, Barrett FS, MacLean KA, Jesse R, Johnson MW, Griffiths RR. Survey study of challenging experiences after ingesting psilocybin mushrooms: Acute and enduring positive and negative consequences. J Psychopharmacol. 2016 Dec;30(12):1268-1278. doi: 10.1177/0269881116662634. Epub 2016 Aug 30. PMID 27578767
- [Background] Yaden DB, Potash JB, Griffiths RR. Preparing for the Bursting of the Psychedelic Hype Bubble. JAMA Psychiatry. 2022 Oct 1;79(10):943-944. doi: 10.1001/jamapsychiatry.2022.2546. PMID 36044208
- [Background] Glynos NG, Pierce J, Davis AK, McAfee J, Boehnke KF. Knowledge, Perceptions, and Use of Psychedelics among Individuals with Fibromyalgia. J Psychoactive Drugs. 2023 Jan-Mar;55(1):73-84. doi: 10.1080/02791072.2021.2022817. Epub 2022 Jan 10. PMID 35001856
- [Background] Ramachandran V, Chunharas C, Marcus Z, Furnish T, Lin A. Relief from intractable phantom pain by combining psilocybin and mirror visual-feedback (MVF). Neurocase. 2018 Apr;24(2):105-110. doi: 10.1080/13554794.2018.1468469. Epub 2018 May 15. PMID 29764303
- [Background] Bornemann J, Close JB, Spriggs MJ, Carhart-Harris R, Roseman L. Self-Medication for Chronic Pain Using Classic Psychedelics: A Qualitative Investigation to Inform Future Research. Front Psychiatry. 2021 Nov 12;12:735427. doi: 10.3389/fpsyt.2021.735427. eCollection 2021. PMID 34867525
- [Background] Bondesson E, Larrosa Pardo F, Stigmar K, Ringqvist A, Petersson IF, Joud A, Schelin MEC. Comorbidity between pain and mental illness - Evidence of a bidirectional relationship. Eur J Pain. 2018 Aug;22(7):1304-1311. doi: 10.1002/ejp.1218. Epub 2018 Apr 16. PMID 29577509
- [Background] Kuner R, Flor H. Structural plasticity and reorganisation in chronic pain. Nat Rev Neurosci. 2017 Jan 20;18(2):113. doi: 10.1038/nrn.2017.5. No abstract available. PMID 28704354
- [Background] Carhart-Harris RL, Leech R, Hellyer PJ, Shanahan M, Feilding A, Tagliazucchi E, Chialvo DR, Nutt D. The entropic brain: a theory of conscious states informed by neuroimaging research with psychedelic drugs. Front Hum Neurosci. 2014 Feb 3;8:20. doi: 10.3389/fnhum.2014.00020. eCollection 2014. PMID 24550805
- [Background] Castellanos JP, Woolley C, Bruno KA, Zeidan F, Halberstadt A, Furnish T. Chronic pain and psychedelics: a review and proposed mechanism of action. Reg Anesth Pain Med. 2020 Jul;45(7):486-494. doi: 10.1136/rapm-2020-101273. Epub 2020 May 4. PMID 32371500
- [Background] MacCallum CA, Lo LA, Pistawka CA, Deol JK. Therapeutic use of psilocybin: Practical considerations for dosing and administration. Front Psychiatry. 2022 Dec 1;13:1040217. doi: 10.3389/fpsyt.2022.1040217. eCollection 2022. PMID 36532184